CLINICAL TRIAL: NCT06610786
Title: The Use of FCSB in Medium-complex RRD - a Safety and Efficacy Evaluation
Brief Title: Foldable Capsular Scleral Buckling Versus Vitrectomy in Medium-complex Rhegmatogenous Retinal Detachment Treatment
Acronym: FCSB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCSB
Record Dates: First submitted 2024-09-11; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Rhegmatogenous Retinal Detachment
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FCSB (Experimental): Using foldable capsular scleral buckle surgery to treat primary rhegmatogenous retinal detachment (RRD) of medium complexity
  Interventions: Procedure: foldable capsular scleral buckling
- PPV (Active Comparator): Using pars plana vitrectomy to treat primary rhegmatogenous retinal detachment (RRD) of medium complexity
  Interventions: Procedure: vitrectomy

INTERVENTIONS:
Procedure: foldable capsular scleral buckling — Using foldable capsular vitreous body as a novel scleral buckle material to treat the primary rhegmatogenous retinal detachment (RRD) of medium complexity
  Arms: FCSB
Procedure: vitrectomy — Using vitrectomy to treat primary rhegmatogenous retinal detachment (RRD) of medium complexity.
  Arms: PPV

SUMMARY:
The objective of the study is to evaluate:

1. Safety and efficacy of a novel foldable capsular scleral buckle (FCSB) in scleral buckling for primary rhegmatogenous retinal detachment (RRD) of medium complexity.
2. Comparison between FCSB and pars plana vitrectomy in therapeutic effects and complications in the treatment of primary RRD of medium complexity.

DETAILED DESCRIPTION:
Pars plana vitrectomy (PPV) and scleral buckling (SB) are major choices in treating rhegmatogenous retinal detachment (RRD) of medium complexity. PPV is more prevailed since it improved internal search for breaks and elimination of vitreous traction. SB has unmatched advantages over PPV such as earlier rehabilitation, free from prolonged positioning, less complicated cataract or glaucoma. The novel foldable capsular scleral buckle (FCSB) can create a big bulge by pressing on the sclera and seal the break in bullous RRD without scleral drainage. In the study, differences of anatomic and functional results between PPV and FCSB in treating primary RRD of medium complexity are evaluated.

ELIGIBILITY:
Inclusion Criteria:

One or more retinal holes which cannot be treated sufficiently with a single silicon sponge or silicone band (e.g. large holes, multiple holes, multiple holes of varying anterior-posterior localisation, massive traction)

Exclusion Criteria

1. simple rhegmatogenous retinal detachment which can be treated with a single silicon sponge or silicone band (e.g. single holes, no traction, limit retinal detachment)
2. Complicated RRD, including macular hole within the arcade, PVR C or D, severe cataract, severe vitreous hemorrhage, unclear macular hole,
3. Combined with other eye diseases that affect vision prognosis.
4. History of other eye surgeries including cataract surgery.
5. Presence of systemic diseases that may affect postoperative observation and follow-up.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
anatomic success rate | From enrollment to the end of treatment at 6 months
  The success rate of retinal reattachment
metamorphopsia | From enrollment to the end of treatment at 6 months
  metamorphopsia is measured by M chart
Visual Results | From enrollment to the end of treatment at 6 months
  Best-Corrected Visual Acuity, and is measured by Snellen Chart, EDTRS Chart and charts designed for people with low vision

SECONDARY OUTCOMES:
The number of surgeries that achieved successful final retinal reattachment | From enrollment to the end of treatment at 6 months
  The number of surgeries the patient undergoes to achieve final retinal reattachment
Surgical Complications | From enrollment to the end of treatment at 6 months
  Surgical Complications, included EOM dysfunction，Choroidal detachment，Clinical CME，Macular pucker，Postoperative IOP >21 mmHg with medications

CONTACTS AND LOCATIONS:
Locations (1):
- EyeEntFudan, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No